CLINICAL TRIAL: NCT06735027
Title: A Randomized Comparative Cohort Study of the Use of Intra-articular Corticosteroid Injection Compared to Suprascapular Nerve Block for Treatment of Shoulder Pain
Brief Title: Corticosteroid Injection Versus Nerve Block
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ORTHOSURG-2024-33106
Record Dates: First submitted 2024-12-03; First posted 2024-12-16 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Glenohumeral Arthritis; Rotator Cuff Arthropathy
Keywords: osteoarthritis; glenohumeral arthritis; rotator cuff arthropathy; corticosteroid injection; suprascapular nerve block
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Two study arms, with each arm receiving one of two interventions: corticosteroid shoulder injection or suprascapular nerve block
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intraarticular methylprednisolone acetate injection (IACI) (Experimental): Patients with glenohumeral osteoarthritis, rheumatoid arthritis, or rotator cuff arthropathy who are poor surgical candidates or who are not interested in pursuing surgery randomized to intraarticular corticosteroid injection (IACI).
  Interventions: Other: intraarticular corticosteroid injection (IACI)
- suprascapular nerve block (SSNB) with bupivacaine and triamcinolone (Experimental): Patients with glenohumeral osteoarthritis, rheumatoid arthritis, or rotator cuff arthropathy who are poor surgical candidates or who are not interested in pursuing surgery randomized to suprascapular nerve block (SSNB)
  Interventions: Other: suprascapular nerve block (SSNB)

INTERVENTIONS:
Other: intraarticular corticosteroid injection (IACI) — The patient will be in a seated position. Correct patient, laterality, and procedure will be performed during the timeout. Ultrasound guidance will be used to identify the glenohumeral joint. The injection site will then be disinfected with an alcohol wipe. A 21, 22, or 23-gauge needle (depending on provider preference) will be advanced into the glenohumeral joint under direct ultrasound visualization. After entry into the glenohumeral joint, a negative aspiration will be performed. At that time, up to 1 mL of 40mg/mL methylprednisolone acetate will be injected be injected into the joint space.
  Arms: intraarticular methylprednisolone acetate injection (IACI)
Other: suprascapular nerve block (SSNB) — The patient will be in a seated position. Correct patient, laterality, and procedure will be performed during the timeout. Ultrasound guidance will be used to identify the suprascapular nerve in its path at the suprascapular notch. After disinfection of the injection site with alcohol, anatomic landmarks for SSNB as described by Dangoisse et al. [10] will be marked with a marking pen. Ultrasound will be utilized to guide the tip of a 21, 22, or 23 gauge (depending on provider preference) needle to the floor of the suprascapular fossa while avoiding neurovascular structures. At that time, a mixture of up to 10 mL of 0.5% bupivacaine and 20 mg triamcinolone will be slowly injected to fill the fascial contents of the suprascapular fossa under direct ultrasound guidance.
  Arms: suprascapular nerve block (SSNB) with bupivacaine and triamcinolone

SUMMARY:
The purpose of this study is to evaluate conservative pain relief measures for patients suffering from glenohumeral arthritis or rotator cuff arthropathy. Conservative management of osteoarthritis is often first line treatment, and while a corticosteroid injection is frequently used, suprascapular nerve blocks have not often been described as an analgesic option in this population.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of glenohumeral osteoarthritis, rheumatoid arthritis, or rotator cuff arthropathy who are being offered injection

Exclusion Criteria:

* uncontrolled diabetes (patients will be excluded if no HbA1c within a year or if it is 8 or greater"
* known allergy to steroid or anesthetic
* pregnant women
* prisoners
* patients with diminished capacity to consent to participation
* children under 18 years of age
* non-English speakers

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2027-01-02 (Estimated); Study Completion 2027-01-02 (Estimated)

PRIMARY OUTCOMES:
change in visual analog scale (VAS) for pain | preintervention, 24 hours, 3 days, 1 month, and 3 months postintervention
  a validated continuous scale assessment for pain
single assessment numerical evaluation (SANE) of the shoulder | preintervention, 24 hours, 3 days, 1 month, and 3 months postintervention
  a validated tool providing a numerical score from 0-100 that assess shoulder function as subjectively reported by the subject. A higher score indicates superior shoulder function.
Oxford shoulder score (OSS) | preintervention, 24 hours, 3 days, 1 month, and 3 months postintervention
  a validated patient-reported outcome measure used to assess shoulder pain and functional disability. Possible scores range from 0-48 with higher scores indicating superior better shoulder function.
American shoulder and elbow surgeons (ASES) score | preintervention, 24 hours, 3 days, 1 month, and 3 months postintervention
  a validated survey with possible scores from 0-100 that assesses shoulder function as reported by the subject. A higher score indicates superior shoulder function.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Rao, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States